CLINICAL TRIAL: NCT01957852
Title: Can FloSeal Reduce the Risk of Intra-abdominal Bleeding After Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy Performed for the Treatment of Peritoneal Carcinomatosis ?
Brief Title: FloSeal in CRS and HIPEC
Status: Completed | Type: Observational
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Principal Investigator, Pierre Dubé, Surgical oncologist, Maisonneuve-Rosemont Hospital
Other Study IDs: 13019
Record Dates: First submitted 2013-05-21; First posted 2013-10-08 (Estimated); Last update posted 2015-02-25 (Estimated); Status verified 2015-02

CONDITIONS: Peritoneal Carcinomatosis
MeSH Terms: conditions — Peritoneal Neoplasms | interventions — FloSeal Matrix

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- FloSeal +: Routine use of Floseal during cytoreductive and HIPEC surgery
  Interventions: Other: FloSeal
- FloSeal -: FloSeal not used during CRS and HIPEC procedure

INTERVENTIONS:
Other: FloSeal
  Other Names: gelatin matrix thrombin solution (Baxter)
  Groups: FloSeal +

SUMMARY:
Introduction

Modern treatment of peritoneal carcinomatosis (PC) combines an aggressive cytoreductive surgery (CRS) of all macroscopic disease and hyperthermic intraperitoneal chemotherapy (HIPEC) performed at the time of surgery. It is considered a high risk procedure and post-operative intra-abdominal bleeding is a major issue as it can delay recovery and promote intra-abdominal infections. In most severe cases (10 to 20% of patients), a second surgery to control the bleeding will be necessary. Major causes of bleeding are : radical resection, extensive peritonectomy, length of surgery, massive transfusion and use of HIPEC.

To reduce the risk of intra-abdominal hemorrhage, many strategies have been tried and one of these is the liberal use of FloSeal, but there is no data in this particular field of interest. Over the last 18 months, the investigators have started to use FloSeal in all their cases with large PC and they have observed a dramatic reduction in the rate of reoperation for bleeding and probably secondarily, in the use of blood products, but this has not been measured.

Hypothesis

FloSeal can reduce the risk of bleeding after CRS and HIPEC procedure.

Primary objective

To evaluate if the use of FloSeal can reduce the risk of reoperation after CRS and HIPEC procedure in the treatment of PC.

Secondary objectives

* To evaluate if the use of FloSeal can reduce operative blood loss.
* To evaluate if the use of FloSeal can reduce the need of blood products after CRS and HIPEC procedure.
* To evaluate if the use of FloSeal can have an impact on other common surgical complications (which can be indirectly bleeding related).
* To evaluate if the use of FloSeal can have an impact on length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients older than 18 year old
* All cases of PC regardless of primary tumour (colorectal carcinoma, peritoneal mesothelioma, appendiceal carcinoma etc.)

Exclusion Criteria:

* Prophylactic HIPEC
* Peritoneal Carcinomatosis Index (PCI) < 5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with peritoneal carcinomatosis (PC) of any cause followed at Hôpital Maisonneuve-Rosemont and undergoing Cytoreductive and HIPEC surgery
Sampling Method: Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2008-01; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Reoperation rate for intra-abdominal bleeding after CRS and HIPEC | postoperative day O to hospital discharge (an expected average of 3 weeks after surgery)

SECONDARY OUTCOMES:
operative blood loss | Cytoreductive and HIPEC surgery
Blood products use | during cytoreductive and HIPEC surgery and post-operative hospital stay (an expected average of 3 weeks)
  packed red blood cells, fresh frozen plasma, platelets, specific coagulation factors and cryoprecipitates
Hemoglobin rate | at hospital discharge (an expected average of 3 weeks)
Non-hemorrhagic complications | postoperative day 0 to hospital discharge (an expected average of 3 weeks after surgery)
  According to the Dindo-Clavien postoperative complications classification
Length of hospital stay | postoperative day 0 to hospital discharge (an expected average of 3 weeks after surgery)
  Hospital discharge is defined in our study as medical discharge

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Dubé, Principal Investigator — Maisonneuve-Rosemont Hospital
Locations (1):
- Hôpital Maisonneuve-Rosemont, Montreal, Quebec, Canada